CLINICAL TRIAL: NCT03780582
Title: Evaluation of Use of Diagnostic AI for Lung Cancer in Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ensemble Group Holdings, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: EN-122018
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probabilistic Classification (Experimental): Radiologists see a "score" from 1-100 that represents the AI's prediction of whether the CT-scan comes from a patient with cancer or not before beginning their analysis of the scan.
  Interventions: Behavioral: AI-human interaction
- Classification Plus Detection (Experimental): Radiologists see a "score" from 1-100 that represents the AI's prediction of whether the CT-scan comes from a patient with cancer or not before beginning their analysis of the scan. They also see ROIs identified by the AI that represent lung nodules.
  Interventions: Behavioral: AI-human interaction
- Classification With Delayed Detection (Experimental): Radiologists see a "score" from 1-100 that represents the AI's prediction of whether the CT-scan comes from a patient with cancer or not before beginning their analysis of the scan. After identifying their own ROIs, the radiologist then can see ROIs identified by the AI that represent lung nodules before making final decisions.
  Interventions: Behavioral: AI-human interaction

INTERVENTIONS:
Behavioral: AI-human interaction — Exploring what kinds of AI-human interaction improve radiologists detection accuracy.

SUMMARY:
This study investigates ways of improving radiologists performance of the classification of CT-scans as cancerous or non-cancerous. Participants interact with an AI to classify CT-scans under three different conditions.

DETAILED DESCRIPTION:
The three conditions are as follows: "probabilistic classification", where the radiologist diagnoses scans using an AI cancer likelihood score; "classification plus detection", where the radiologist see detecting lung nodules in addition to the AI's probabilistic classification score before making her own examination of the CT-scan; and "classification with delayed detection", where the radiologist identifies regions of interest independently of the AI and then sees the AI's detected ROIs.

ELIGIBILITY:
Inclusion Criteria:

* The participant performs radiology screenings professionally

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Classification accuracy | up to 4 months after initiation of evaluation of the test set
  This compares radiologists' classifications with the ground truth in the tested cases.

SECONDARY OUTCOMES:
detection concordance | up to 4 months after initiation of evaluation of the test set
  Evaluation of concordance between radiologists in the tested cases in detection of lung nodules > 4 mm

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided